CLINICAL TRIAL: NCT03650829
Title: IVF Offspring Born in Guangzhou Cohort Study
Brief Title: IVF Offspring Born in Guangzhou
Acronym: IVF-BIG
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2018080103
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: ART; Offspring, Adult; Genetics; Host and Microbiome; Neurodevelopment
Keywords: ART; Offspring; Development; Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine and stool. At delivery: cord, cord blood and placenta. During Infancy：dry blood spot, stool and blood. During childhood:blood, buccal swab and stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The IVF Offspring Born in Guangzhou Cohort Study (IVF-BIG) was established to investigate the short- and long-term effects of exposure in early life on the health of mothers and offspring in Guangzhou, China. Data are collected regarding assisted reproductive technology (ART), environmental, occupational and lifestyle exposures as well as health outcomes in their later life. Biological samples including blood and tissue samples are also collected from participants.

DETAILED DESCRIPTION:
It has been 40 years since the first IVF baby born in the world. The effects of hormonal drugs used on women and health of IVF offspring have always been concerned in the reproductive field and in public. With the increase of the prevalence of infertility and development of ART, China is facing a IVF babies boom. It has been reported that ART was associated with higher risk of cancers among women undergoing treatment of ART, and an increased incidence of autism and noncommunicable chronic diseases, such as obesity, among IVF offspring. Epigenetics is documented as one of the possible mechanisms, while answers remain to be explored. A birth cohort would provide an opportunity to examine the short- and long-term effects of ART exposure on health consequences of the mothers and babies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with <20 weeks of gestation
* Pregnant women intended to eventually deliver in Guangzhou Women and Children's Medical Center
* Permanent residents or families intended to remain in Guangzhou with their child for ≥3 years
* Pregnant women conceived by assited reproductive technology

Exclusion Criteria:

• None

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Mothers conceived by ART in the BIGCS
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Intelligence quotient of offspring | At age of 6 years old
  Assessed using Wechsler's Intelligence Scale of Children (WISC) including verbal test and performance test.Intelligence quotient ranges from 40 to 160, in which under 70 is defined as mental retardation

SECONDARY OUTCOMES:
Prevalence of gestational diabetes, pregnancy induced hypertension, and cesarean section | From 20 weeks of gestation to delivery
  Assessed by self-reported time of onset and electronic medical records
Prevalence of stillbirth, preterm birth, small for gestational age, large for gestational age and birth defect | At delivery
  Assesed by electronic records
Neurodevelopment at early childhood | At age of 1 year old
  Assessed using Gesell Developmental Schedules, including five items of adaptive, gross motor, fine motor, language, and social function
Epegenetic profiles of offspring | At age of 1 year, 6 years, 12years and 18 years old
  Profiling DNA methylation and histone acetylation etc., using blood samples
Changes of body composition and bone density during early childhood | At age of 3 years,6 years, 12 years and 18 years old
  Assessed using Dual Energy X-Ray Absorptiometry
Height changes during early childhood | At birth, age of 6 weeks, 6 months, 1 year and 3 years old
  Height changes from birth, to age of 6 weeks, 6 months, 1 year and 3 years old
Weight changes during early childhood | At birth, age of 6 weeks, 6 months, 1 year and 3 years old
  Weight changes from birth, to age of 6 weeks, 6 months, 1 year and 3 years old
Change of intestinal flora during early childhood | At age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
  Assessed by analyses of stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694
- See also: Related website — http://www.bigcs.com.cn